CLINICAL TRIAL: NCT00171405
Title: A 4 Month Extension to a 12 Month, Randomized, Open-label, Multicenter, Study to Assess the Long-term Safety of Aliskiren 150 mg Alone and 300 mg Alone or With the Optional Addition of Hydrochlorothiazide (12.5 mg or 25 mg) in Patients With Essential Hypertension
Brief Title: A Clinical Study to Evaluate the Long-term Safety (12 Months) of the Combination of Aliskiren 300 mg and Hydrochlorothiazide 25 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A2302E1
Record Dates: First submitted 2005-08-24; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: hypertension; aliskiren; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
The purpose of this study is to collect the long-term (12 months) safety data on aliskiren 300 mg when taken in combination with HCTZ 25 mg.

ELIGIBILITY:
Inclusion Criteria:

1. their successful completion of the CSPP100A2302 core study with at least eight months combination treatment of aliskiren 300 mg and HCTZ 25 mg, i.e., patients who received aliskiren 300 mg and HCTZ 25 mg at Month 4 of the core study and complete the core study.
2. absence of ongoing severe adverse events at Visit 10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Assessment of safety through reporting of adverse events and serious adverse events, including deaths, following a 12 month study

SECONDARY OUTCOMES:
Change from baseline (following a 12 month study) in mean sitting diastolic blood pressure after 4 months
Change from baseline (following a 12 month study) in mean sitting systolic blood pressure after 4 months
Change from baseline (following a 12 month study) in mean standing blood pressure after 4 months
Diastolic blood pressure less than 90 mmHg or 10 mmHg or greater change from baseline
Blood pressure less than 140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Investigative Site, East Hanover, New Jersey, United States
- Investigative Site, Deurne, Belgium
- Investigative Site, Ste-Fov, Canada
- Investigative Site, Krassel, Germany
- Investigative Site, Broni, Italy
- Investigative Site, Rotterdam, Netherlands
- Investigative Site, Lima, Peru
- Investigative Site, Moscow, Russia
- Investigative Site, Basel, Switzerland
- Investigative Site, London, United Kingdom

REFERENCES:
- [Result] Sica D, Gradman AH, Lederballe O, Kolloch RE, Zhang J, Keefe DL. Long-term safety and tolerability of the oral direct renin inhibitor aliskiren with optional add-on hydrochlorothiazide in patients with hypertension: a randomized, open-label, parallel-group, multicentre, dose-escalation study with an extension phase. Clin Drug Investig. 2011 Dec 1;31(12):825-37. doi: 10.1007/BF03256921. PMID 22035463